CLINICAL TRIAL: NCT00664157
Title: Facial Expression Recognition of Emotion and Categorization of Emotional Words in Parkinson's Disease. Impact of L-Dopa and Deep Brain Stimulation of Subthalamic Nucleus .
Brief Title: Facial Expression Recognition of Emotion and Categorization of Emotional Words in Parkinson's Disease. Impact of L-Dopa and Deep Brain Stimulation of Subthalamic Nucleus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Pr Durif, CHU Clermont-Ferrand
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: CHU-0033; RBHP 2007 Durif
Record Dates: First submitted 2008-04-21; First posted 2008-04-22 (Estimated); Last update posted 2011-01-19 (Estimated); Status verified 2011-01

CONDITIONS: Idiopathic Parkinson's Disease
Keywords: Idiopathic Parkinson's disease; L-Dopa; Deep Brain stimulation; Facial expression recognition of emotion; Frequency levels; Automatic and voluntary information treatment; Patient with an Idiopathic Parkinson's disease
MeSH Terms: conditions — Parkinson Disease

ARMS (1):
- 2 (Other): 40 patients with an idiopathic Parkinson's disease and 40 healthy paired volunteers (control group)
  Interventions: Behavioral: Facial expression recognition of emotion

INTERVENTIONS:
Behavioral: Facial expression recognition of emotion — Facial expression recognition test Lexical decisiontest
Behavioral: Facial expression recognition of emotion — Facial expression recognition test Lexical decision test

SUMMARY:
Parkinson'disease is a neurodegenerative disorder characterised by bradykinesia, rigidity, rest tremor and postural instability. Dopaminergic therapy such as L-Dopa and dopamine agonists usually leads to a dramatic improvement of symptoms, but disease progression nevertheless remains inevitable. Bilateral Deep brain stimulation in subthalamic nucleus is now considered the gold standard surgical treatment.

Parkinson'disease mainly affects the nigrostriatal dopaminergic system which is linked to the limbic system and could be responsible of a specific trouble in the recognition in some facial expression.

We hypothesise that patients with Parkinson'disease present a dysfunction of voluntary and automatic treatment of emotional information.

The main purpose of this study is to show if patients with Parkinson'disease present a lack of specific facial expression recognition of emotion and determinate more precisely if this alteration involves the cortical way (high frequency way) or the under cortical way (low frequency way).

We also examine the role of L-Dopa and the deep brain stimulation on emotion perception

DETAILED DESCRIPTION:
40 patients with an Idiopathic Parkinson's disease divided in two groups :

* 20 patients evaluated before surgery and 6 month after surgery
* 20 patients only evaluated after surgery.

  40 paired healthy volunteers

  1) Study progress (patients):

Inclusion visit :

Neurological evaluations .

Neuropsychological evaluations : MMS, MADRS, MATTIS, BREF, Wisconsin test, Apathy test, Benton….

Ophthalmic visit : VISTECH

Protocol :

1. for patients evaluated before surgery Facial expression recognition test Lexical decision test Made in two conditions : without the treatment (Med OFF) and one hour after the L-Dopa administration (MED ON)
2. for patients evaluated after surgery Facial expression recognition test Lexical decision test Made in four conditions

   * Without stimulation (STIM OFF) and medication (MED OFF)
   * MED OFF and STIM ON
   * MED ON and STIM OFF
   * MED ON and STIM ON

     2) Study progress (healthy volunteers): Ophthalmic visit MMS Facial expression recognition test Lexical decision test

ELIGIBILITY:
Inclusion Criteria:

* Age : 30-75 years
* Patient with an idiopathic Parkinson's disease according to the criteria of the "Parkinson's Disease Society Brain Bank" (Hughes et al., 1992)
* Patient treated with a deep brain stimulation according to the French consensus conference of treatment of Parkinson's disease (Consensus Conference Proceeding, 2000)
* Effect of the stimulation 50%
* Affiliation to social security
* Agreement of patients

Exclusion Criteria:

* Patients suffering of an atypical Parkinson syndrome
* Patients with severe tremor before surgery
* Patients with a vision contrast altered.
* Patients who do not understand the words associated with an emotion
* Pregnant women
* Person who participate to an other study

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2007-09; Primary Completion 2008-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Facial expression recognition test | % of exact responses

SECONDARY OUTCOMES:
Lexical decision test | The time to respond

CONTACTS AND LOCATIONS:
Overall Officials: Franck Durif, PUPH, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU, Clermont-Ferrand, France